CLINICAL TRIAL: NCT06516796
Title: Omitting of Lymphadenectomy is Acceptable for Lung Cancer Smaller Than 6 mm in Solid Size
Status: Completed | Type: Observational
Sponsor: Liang Chen (Other)
Responsible Party: Sponsor-Investigator, Liang Chen, Director, Head of Thoracic Surgery, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Other Study IDs: 2022-SR-760
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Sublobar resection; Non-small cell lung cancer; No lymphadenectomy; Solid size
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- sublobar resection without lymphadenectomy: Patients received sublobar resection but had no lymphadenectomy
  Interventions: Other: No intervention
- sublobar resection with lymphadenectomy: Patients received sublobar resection plus lymphadenectomy
  Interventions: Other: No intervention
- lobectomy plus lymphadenectomy: Patients received lobectomy plus lymphadenectomy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients were retrospectively screened.

SUMMARY:
Many studies suggested that selective lymph node sampling was acceptable for specific non-small cell lung cancer (NSCLC). This study aimed to evaluate the acceptability of omitting of lymphadenectomy for selected NSCLC.

Patients with small-sized (≤2 cm) NSCLC who underwent surgical resection between 2009 and 2022 were retrospectively screened.

DETAILED DESCRIPTION:
Many studies suggested that selective lymph node sampling was acceptable for specific non-small cell lung cancer (NSCLC). This study aimed to evaluate the acceptability of omitting of lymphadenectomy for selected NSCLC.

Patients with small-sized (≤2 cm) NSCLC who underwent surgical resection between 2009 and 2022 were retrospectively screened. The characteristics of patients with nodal metastasis were demonstrated. For selected patients, the perioperative and long-term outcomes of patients with and without lymphadenectomy were compared. Log-rank test and Cox regression analysis were adopted for prognostic evaluation.

A total of 2713 NSCLC patients were enrolled, and 75 of them (2.76%) had nodal involvement. None of patients with pure ground glass opacity (0/945) had nodal metastasis, while 14 patients with part-solid (14/1260, 1.11%) and 61 patients with solid nodules (61/508, 12.01%) had nodal involvement. Patients with nodal metastasis had a minimum solid size of 6 mm. NSCLC with solid components < 6 mm (n=1588) had no nodal metastasis. Of them, 339 patients underwent sublobar resection without lymphadenectomy (SRN0), 1056 subjects received sublobar resection with lymphadenectomy (SRN1), and 190 patients received lobectomy plus lymphadenectomy (LRN1). Patients with SRN0 had a shorter operating time, less volume of drainage, a lower incidence of chylothorax (0 vs. 0.6% vs. 2.1%, P=0.012) and air leakage, as well as a shorter postoperative hospitalization (3 vs. 4 vs. 4 days, P<0.001) than those with SRN1 or LRN1. During a median follow-up of 61 months, no patient with SRN0 was dead or tumor recurrent. The 5-year recurrence-free survival was 100%, 99.2% and 98.5% for patients with SRN0, SRN1 and LRN1, respectively (P=0.370).

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed non-small cell lung cancer (NSCLC)
* the maximum tumor diameter ≤2 cm
* receiving surgical treatment between 2009-2022

Exclusion Criteria:

* non-primary NSCLC;
* with small cell lung cancer components;
* undergoing preoperative neoadjuvant therapies;
* with compromised resection;
* malignant tumor history over the past five years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-small cell lung cancer with a total tumor size within 2 cm
Sampling Method: Non-Probability Sample
Enrollment: 2713 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | OS was defined from the surgical date to the date of death or the date of the last follow-up, whichever came first, assessed up to 14 years.
  OS was defined from the surgical date to the date of death or the date of the last follow-up. defined from the surgical date to the date of death or the date of the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No